CLINICAL TRIAL: NCT01643434
Title: Multicenter Study of Patients With Hypertension Resistant to Patient Identification and Standardization of Therapeutic
Brief Title: Resistant Hypertension Optimal Treatment
Acronym: ReHOT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Eduardo Moacyr Krieger, PI, Instituto do Coracao
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0758/09
Record Dates: First submitted 2012-07-11; First posted 2012-07-18 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension
Keywords: Resistant Hypertension
MeSH Terms: conditions — Hypertension | interventions — Spironolactone; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone
- Clonidine (Active Comparator)
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Spironolactone — Spironolactone (titrating dose from 12.5 to 50mg SID)
  Arms: Spironolactone
Drug: Clonidine — Clonidine (titrating dose from 0.100-0.300mg BID)
  Arms: Clonidine

SUMMARY:
Resistant hypertension (ReHy) is an emerging clinical and public health problem which tends to increase because populations are living longer and there is a growing global epidemic of obesity, diabetes and sleep apnea. It is also tempting to speculate that the excessive dietary salt ingestion reported in many countries can contribute substantially to the risk of ReHy development. ReHy is defined as persistent high blood pressure (above the target goal) in spite of the use of at least 3 antihypertensive agents of different classes, one of them must being diuretics.

Data regarding the exact prevalence of ReHy are very limited. In addition, little data is available about 3-drug combinations but a simplified treatment algorithm has demonstrated that a combination of a diuretic plus an angiotensin-converting enzyme inhibitors (ACEi) or an angiotensin-receptor blocker (ARB) plus diuretic, adding a calcium channel blocker when necessary, controlled 64% of hypertensive patients and, in addition, was even more efficient than the current guideline-based management. By contrast, the fourth drug to be added-on the triple regimen is still controversial and guided by empirical choices or personal preferences. Recent studies suggest the emerging role of spironolactone as the "first-line" fourth drug for treating resistant hypertension. Conversely, because of the pathophysiological rationale, others have proposed the use of β-blockers or even centrally acting agents for managing the sympathetic hyperactivity. The present concerns about the limited blood pressure reducing effect of β-blockers, especially in elderly people, the potent effect of centrally acting agents and our personal experience are pointing to clonidine as the fourth drug to be added-on to a multidrug combination for reaching optimal blood pressure in patients with ReHy. Nevertheless, no studies have been performed comparing, head-to-head, which one is the best fourth drug (spironolactone or clonidine) to be added-on to a common used multidrug combination in order to treat this condition.

Therefore, the principal objectives of the ReHOT Trial are to assess prospectively: (1) the prevalence of ReHy in a cohort of outpatients with stage II hypertension; (2) the effect of spironolactone on blood pressure, in comparison to clonidine, when added to a multidrug combination consisting of chlorthalidone plus ACEi (or ARB) plus amlodipine, all of 3 up-titrated to the highest dose; (3) the role of measuring sympathetic nervous system activity and renin-angiotensin-aldosterone activity on predicting the response of blood pressure to spironolactone and clonidine.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged between 18 and 75
2. With systolic blood pressure> 160 mmHg and <220mmHg and / or diastolic> 100 mmHg in the sitting position and according to Brazilian Guidelines on Hypertension (perform steps by obtaining two consecutive measurements differing by less than 4 mmHg between them, calibrated using a sphygmomanometer)
3. Patient regularly enrolled in participating center

Exclusion criteria

1. Systolic blood pressure> 220 mmHg
2. Patients with cardiovascular events (stroke, AMI, etc.). or cardiovascular procedures with less than 6 months of evolution
3. Renal stages IV and V (glomerular20 filtration estimated by MDRD formula <30 ml / min; where MDRD = 186 x (S_Cr) -1.154 x (age) -0.203 x (0.742 if fem.) x (1.210 if Afro-amer. ))
4. Heart failure class III and IV
5. History of malignant disease with life expectancy < 2 years
6. Alcoholism
7. Psychiatric illnesses that prevent compliance with the Protocol
8. Women of childbearing age who are not in use of effective contraception
9. Pregnancy
10. Arrhythmias, valvular heart disease, AV block 2 and 3 degrees without MP
11. Hepatic impairment
12. Patients with a history of hypersensitivity to any of the drugs under study
13. Examination of the fundus: Grade III and Grade IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (mmHg) | Patients willl be followed for an expected average of 3 months
  Compare the effect of spironolactone on blood pressure vs. clonidine, when added to a multidrug combination consisting of chlorthalidone plus ACEi (or ARB) plus amlodipine, all of 3 up-titrated to the highest dose;

SECONDARY OUTCOMES:
Sympathetic nervous system and renin-angiotensin-aldosterone activity | At baseline and at the end of the randomization (3 months)
  Compare the role of measuring sympathetic nervous system activity and renin-angiotensin-aldosterone activity on predicting the response of blood pressure to spironolactone and clonidine.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M. Krieger, Doctor, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Krieger EM, Drager LF, Giorgi DMA, Pereira AC, Barreto-Filho JAS, Nogueira AR, Mill JG, Lotufo PA, Amodeo C, Batista MC, Bodanese LC, Carvalho ACC, Castro I, Chaves H, Costa EAS, Feitosa GS, Franco RJS, Fuchs FD, Guimaraes AC, Jardim PC, Machado CA, Magalhaes ME, Mion D Jr, Nascimento RM, Nobre F, Nobrega AC, Ribeiro ALP, Rodrigues-Sobrinho CR, Sanjuliani AF, Teixeira MDCB, Krieger JE; ReHOT Investigators. Spironolactone Versus Clonidine as a Fourth-Drug Therapy for Resistant Hypertension: The ReHOT Randomized Study (Resistant Hypertension Optimal Treatment). Hypertension. 2018 Apr;71(4):681-690. doi: 10.1161/HYPERTENSIONAHA.117.10662. Epub 2018 Feb 20. PMID 29463627
- [Derived] ReHOT Investigators; Krieger EM, Drager LF, Giorgi DM, Krieger JE, Pereira AC, Barreto-Filho JA, da Rocha Nogueira A, Mill JG. Resistant hypertension optimal treatment trial: a randomized controlled trial. Clin Cardiol. 2014 Jan;37(1):1-6. doi: 10.1002/clc.22228. Epub 2013 Dec 11. PMID 24338935